CLINICAL TRIAL: NCT03436446
Title: Using Social Incentives to Increase Response Rate to Routine Patient Reported Outcome Measurement After Episodic Healthcare Interventions
Brief Title: Role of Social Incentives in PRO Collection
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00086277
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-05

CONDITIONS: Orthopedic Disorder
Keywords: Patient Reported Outcomes (PRO); Social Incentives
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orthopedic Patients: Orthopedic patients will undergo an interview with the research team regarding the framing of various social incentives to promote increased response rates for patient reported outcome measures post-operatively.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Interviews will be conducted with orthopedic patients to review the construction and phrasing of various social incentives aimed at promoting patient reported outcome collection amongst post-operative patients.

SUMMARY:
Value-based healthcare is heavily dependent on the accurate measurement of patient outcomes, both immediately after treatment and at long-term intervals. Patient reported outcomes (PROs) are often the central component of any quality improvement process as they are patient centered, reflect the ultimate objective of the intervention and are endorsed by many professional societies as the preferred physician performance metric. Although high response rates are critical to producing reliable data to support value-based payment models, quality improvement, and stakeholder transparency - especially in arthroscopy in which patients often fare well over time and may be less likely to continue with follow-up - response rates to outcome surveys after initial recovery from treatment are consistently below 50%. Monetary incentives offer only minor improvements in response rates against large increases in already rising costs. Individually tailored social incentives - as grounded in current behavioral economic practice - offer a potential cost-effective solution to this problem in Sports Medicine and arthroscopy.

The investigators predict that well-constructed, personal social incentives will increase response rates for long-term follow-up of episodic care compared to control. The investigators predict these rates will vary depending on the patient demographics and other characteristics.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Orthopedic patient
* 6-24 months post-operative

Exclusion Criteria:

* Non-English speaking

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include post-operative orthopedic patients.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Interview feedback | End of discussion with patient, 15 minutes
  The investigators will use feedback from the interviews to adjust the social incentives.

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Mather III, MD, MBA, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No